CLINICAL TRIAL: NCT05909358
Title: A Phase I/II Randomized Placebo Controlled Trial to Evaluate the Safety and Immunogenicity of Sudan Ebolavirus Vaccines in Uganda
Brief Title: Solidarity/Tokomeza Ebola Trial
Acronym: TOKOMEZA
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Makerere University Lung Institute (Unknown); MRC/UVRI and LSHTM Uganda Research Unit (Other); Makerere University Walter Reed Program (Unknown); Epicentre (Other); Uganda Virus Research Institute-International Aids Vaccine Initiative (Unknown); Ministry of Health, Uganda (Other Government)
Responsible Party: Principal Investigator, Bruce J Kirenga, Prof, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TOKOMEZA PLUS
Record Dates: First submitted 2023-05-30; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Sudan Ebola Virus Vaccines

STUDY DESIGN:
Intervention Model Description: A phase I/II double blind randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinding to be done
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Candidate vaccine 1 (Experimental): One injection of cAd3 will be administered to the study participants at enrollment. The participants will be monitored for 30 minutes after receipt of the vaccine and thereafter follow up done at different time points up to 72 months.
  Interventions: Biological: CAd3
- Candidate vaccine 2 (Experimental): One injection of chAdOx1 will be administered to the study participants at enrollment. The participants will be monitored for 30 minutes after receipt of the vaccine and thereafter follow up done at different time points up to 72 months.
  Interventions: Biological: ChAdox1
- Candidate vaccine 3 (Experimental): One injection of rVSV-SUDV will be administered to the study participants at enrollment. The participants will be monitored for 30 minutes after receipt of the vaccine and thereafter follow up done at different time points up to 72 months.
  Interventions: Biological: rVSV-SUDV
- Control (Placebo Comparator): One injection of placebo will be administered to the study participants at enrollment. The participants will be monitored for 30 minutes after receipt of the vaccine and thereafter follow up done at different time points up to 72 months.
  Interventions: Other: Control

INTERVENTIONS:
Biological: CAd3 — CAd3 candidate vaccine which is one of the investigational products
  Arms: Candidate vaccine 1
Biological: ChAdox1 — ChAdox1 candidate vaccine which is one of the investigational products
  Arms: Candidate vaccine 2
Biological: rVSV-SUDV — rVSV-SUDV candidate vaccine which is one of the investigational products
  Arms: Candidate vaccine 3
Other: Control — Placebo
  Arms: Control

SUMMARY:
The TokomezaPlus Ebola trial is a phase I/II double blind randomised clinical trial designed to assess the safety and immunogenicity of candidate SUDV vaccines in Uganda during the inter outbreak period. Uganda is prone to Ebola virus disease outbreaks especially those caused by the Ebola Sudan (SUDV) species. TokomezaPlus Ebola Vaccine trial protocol has two main components: a) Safety b) Immunogenicity and is designed to create a living protocol that will be used to study the safety and immunogenicity of SUDV-candidate vaccines in the East African EVD-prone countries.

DETAILED DESCRIPTION:
The Sudan ebolavirus and the Zaire ebolavirus are classified as different species, and vaccines and monoclonal antibodies that are effective against Zaire ebolavirus disease are unlikely to be of any use against SUVD. But, the epidemiology of SUVD is thought to be similar to that of Zaire ebolavirus disease.

There is an urgent need to test the safety and immunogenicity of the candidate vaccine(s) developed against Sudan ebolavirus. Once safety and immunogenicity (including extended immunogenicity) have been proven, these vaccines could be deployed for future outbreaks as part of the response.

OBJECTIVES Phase 1 Objectives

1. To determine the safety of rVSV-SUDV candidate SUDV vaccine among healthy volunteers
2. To determine the immunogenicity of rVSV-SUDV candidate SUDV vaccine

Phase 2 Primary objectives

1. To determine the safety of ChAdox1, CAd3 and rVSV-SUDV candidate SUDV vaccine(s) among healthy volunteers and persons with stable comorbidities.
2. To determine the immunogenicity of the three candidate SUDV vaccines.

Secondary objectives

1. To determine the durability of SUDV-specific induced immune responses following vaccination with ChAdox1, CAd3 and rVSV-SUDV candidate SUDV vaccine(s).
2. To determine the factors associated with vaccine-induced immune responses.
3. To determine the putative cross reactivity & protection exerted by the SUDV vaccine candidates against other ebolaviruses (e. g. Bundibugyo ebolavirus (BUDV) and EBOV).

Exploratory objectives

1. To determine the effect of SUDV vaccines on host gene expression
2. To determine the T and B cell specific responses and immune profiling in response to vaccination
3. To determine the effect of SUDV vaccines on the host metabolome
4. To determine the effect of SUDV vaccines on host immune responses

END POINTS

Primary Endpoints

1. Number of solicited, unsolicited adverse and serious adverse events that are determined as possibly, probably and definitely related to the investigational products.
2. Binding antibody titres, neutralization activity and cell mediated immune responses.

Secondary Endpoints

1. Durability of SUDV-specific induced immune responses following vaccination.
2. Factors associated with vaccine-induced immune responses.
3. To determine the putative cross reactivity & protection exerted by the SUDV vaccine candidates against other ebolaviruses (e. g. Bundibugyo ebolavirus (BUDV) and EBOV).

TRIAL PARTICIPANTS This trial will enroll a total 250 healthy, adult volunteers (18-50 years) (150 intervention arm and 100 placebo arm) for the phase I rVSV-SUDV vaccine. The DSMB will review day 28 post vaccination safety data for all the phase I participants and day 56 post vaccination binding antibody IgG and IgM data for 50 participants randomly selected who receive the rVSV SUDV and 10 participants who receive the placebo to make a recommendation regarding proceeding to phase II. Participants enrolled in phase I of the rVSV-SUDV candidate vaccine will contribute data to phase II for this vaccine. For the Phase II trial (ChAdox1, CAd3 and rVSV-SUDV vaccines), 2121 volunteers aged 6 - 65 years will be included (606 for each of the vaccine arms and 303 to placebo). A randomly selected subset of120 participants per vaccine and 50 placebo recipients will participate in extended immunogenicity studies (long term immunogenicity and exploratory studies). 100 participants from each intervention arm participating in extended immunogenicity will randomly be selected to receive a homologous booster 12months post vaccination.

STATISTICAL ANALYSIS The primary analysis is the comparison of occurrence of solicited (within 7 days) and unsolicited adverse events (occurring within 56 days) considered possibly, probably or definitely related to vaccines as well as adverse and SAEs occurring within 24 months' post-vaccination between each candidate vaccine and placebo. AEs will be summarized with counts, percentages, and, when provided, exact 95% CIs will be provided. SAEs will be graded according to DAIDS. The primary analysis for the immunogenicity is the change in serum IgG and IgM titres from baseline to 56days post vaccination.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* Healthy volunteers aged 18-50 years from study communities
* Healthy volunteers with a permanent home address
* Able and willing to complete and provide written informed consent. In case the participant cannot read or write, the procedures must be explained to him/her and informed consent must be witnessed by a literate third party not involved with the conduct of the study
* Participant must pass the informed consent test of understanding (TOU)
* Participant must be healthy in the investigator's clinical judgement on the basis of medical history, physical examination, vital signs and point of care tests (where applicable) performed at screening
* If female of child-bearing potential and heterosexually active, practice of adequate contraception for 28 days prior to injection, negative pregnancy test on the day of vaccination, and agreement to continue adequate contraception until 90 days after vaccination
* Male participants are eligible to participate in the study if they agree to use a male condom during any heterosexual intercourse with a female of childbearing potential until 90 days after vaccination

Phase 2

* Healthy volunteers aged 6 years-65 years from study communities. Individuals with comorbidities assessed as stable will be allowed to participate
* With a permanent home address
* Able and willing to complete and provide written informed consent or assent as applicable. In case the participant cannot read or write, the procedures must be explained to him/her, and informed consent must be witnessed by a literate third party not involved with the conduct of the study.
* Participant must pass the informed consent or assent test of understanding (TOU)
* Participant must be healthy according to the investigator's clinical judgement on the basis of medical history, physical examination, vital signs and point of care tests (where applicable) performed at screening
* If female of child-bearing potential and heterosexually active, practice of adequate contraception for 28 days prior to injection, negative pregnancy test on the day of vaccination, and agreement to continue adequate contraception until 180 days after vaccination
* Male participants are eligible to participate in the study if they agree to abstain from any heterosexual intercourse with a female of childbearing potential or must agree to use a male condom

Exclusion Criteria:

Phase 1

* History of confirmed ebola virus diseases (SUDV, EBOV or BUDV)
* Unwillingness of female participants to use effective contraception
* Participation in an interventional clinical trial within 90 days of participation in this trial
* Prior vaccination with any Ebola vaccine
* Breastfeeding or planning to conceive within 2 months following study vaccination
* Has history of fever (>100.4ºF/38.0ºC) within 48 hours prior to enrolment into the study
* Received systemic corticosteroids exceeding physiologic replacement doses (~5 mg/d prednisone equivalent) within 14 days prior to study entry
* Received any live virus vaccine within 30 days or any non-live virus vaccine within 14 days prior to study entry
* Has a known allergy/sensitivity or contraindication to investigational vaccines or its/their excipients?
* History of malignancy ≤5 years
* Major surgery within the 4 weeks prior to screening or planned major surgery through the course of the study (from screening until completion of the study)
* Presence of any condition that can interfere with the subject's participation for the full duration of the trial.
* HIV positive
* Hepatitis B positive

Phase 2

* History of confirmed SUDV
* Unwillingness of female participants to use effective contraception
* Participation in an interventional clinical trial within 90 days of start of this trial
* Prior vaccination with any Ebola vaccine
* Breastfeeding or planning to conceive within 2 months following study vaccination
* Has history of fever (>100.4ºF/38.0ºC) within 48 hours prior to vaccination
* Received systemic corticosteroids exceeding physiologic replacement doses (~20 mg/d prednisone or equivalent) for 14 days within a month prior to study entry.
* Immunosuppressive medication within 3 months
* Received any live virus vaccine within 30 days or any non-live virus vaccine within 14 days prior to study entry
* Has a known allergy/sensitivity or contraindication to investigational vaccines or its/their excipients?
* History of malignancy ≤5 years
* Major surgery within the 4 weeks prior to screening or planned major surgery through the course of the study (from screening until completion of the study)
* Presence of any condition that can interfere with the subject's participation for the full duration of the trial

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2121 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of solicited, unsolicited adverse and serious adverse events (safety) | 72 months
  The adverse events (AE) and serious adverse events (SAE) will be evaluated to determine the link to the investigational product. They will then be classified as possibly, probably and definitely related to the investigational products
Vaccine-specific antibody concentration (immunogenicity) measured as optical density that will be converted to concentration | 72 months
  The vaccine specific antibody concentration will be assessed through specific laboratory procedures that make use of Nunc Maxisorp flat bottom plates will be coated with Ebola GP in a coating buffer. Heat inactivated serum or plasma from study participants (either diluted and or undiluted) or treated plasma sample from SUDV convalescent individuals (Positive control) or Mouse anti SUDV GP mAb (positive control) will be added to the plates and incubated. The plates will be washed and HRP goat anti-human IgG antibody and or HRP goat anti-human IgM antibody and or HRP goat anti-mouse IgG Fc or HRP goat anti-mouse IgM Fc will be added. The plates will be washed and tetramethylbenzidine (TMB) 1 component microwell peroxidase substrate added. The reaction will be stopped after about 20 minutes with hydrochloric acid. The plate's absorbance will be read at 450 nm and 630 nm. A standard curve/line will be drawn and convert the optical density to concentration
Vaccine specific antibody neutralization capability (immunogenicity) represented as proportion of neutralization | 72 months
  Vero cells will be incubated in Eagles Minimum Essential Medium with fetal bovine serum and penicillin/streptomycin (R10) and maintained at 37°C and 5% CO2 humidified incubator. The cells will be plated onto a 96 well black flat bottomed culture plate.
  Study participant, positive (obtained from SUDV convalescent individuals and pre-treated) and negative controls heat inactivated serum samples will be diluted and mixed with single round infecting recombinant vesicular stomatitis virus expressing SUDV GP and firefly luciferase at room temperature with appropriate controls. The virus and serum sample mixture will be added to the plated vero cells and incubated for up to 24 hours. The virus and serum sample will be removed and vero cells lysed. Luciferase activating reagent will be added and the luminescence will be read using a luminescence plate reader. The proportion of neutralisation will be evaluated using appropriate controls (rVSV without serum).
Vaccine-induced T cell responses (immunogenicity) determined as spot forming units per one million cells. | 72 months
  This will be done as per the standard operating procedures. IFN-γ precoated ELISPOT plates will be washed and blocked using serum. Thawed and rested PBMC will be plated, stimuli (peptides to ebola GP, appropriate positive and negative controls) added and incubated for 12 to 24 hours.
  The plates will be emptied and washed after incubation. Diluted enzyme-conjugate detection IFN-γ antibody will be added and incubated. The plates will be washed & substrate added and allowed to develop for about 20 minutes. The development will be stopped by rinsing the plates in copious amounts of deionised water. The plates will be allowed to air dry in the dark and read using an ELISPOT reader within 12 hours.
  The results will be determined as spot forming units per one million cells

SECONDARY OUTCOMES:
Durability of the immune response measured up to 72 months quantitively by assessing the antibody concentration and qualitatively by assessing the antibody neutralization capacity. Curves will be drawn to represent immune responses against time | 72 months
  Blood samples will be collected at different time points and the immunogenicity assays repeated. Curves will then be drawn to represent how the antibody titers against time

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon reasonable request. The request will be discussed within the trial consortium
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 5 years